CLINICAL TRIAL: NCT05125809
Title: An Operationally Seamless, Randomized Phase 2/3 Study Consisting of a Phase 2 Single-Blind, Dose-Evaluation Phase and a Phase 3 Double-Blind, Placebo-Controlled Phase to Assess the Efficacy and Safety of Setrusumab in Subjects With Osteogenesis Imperfecta
Brief Title: Setrusumab vs Placebo for Osteogenesis Imperfecta
Acronym: Orbit
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UX143-CL301; 2021-006597-23 (EudraCT Number); 2024-510919-29-00 (EU CTIS Number)
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — setrusumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose Setrusumab -> Open-Label (OL) Setrusumab Selected Dose (Experimental): Single-blind setrusumab low dose during Phase 2 followed by open-label setrusumab selected dose
  During treatment and treatment extension periods, participants may receive supplementation with calcium and vitamin D to maintain normal values as directed by the treating physician
  Interventions: Biological: Setrusumab
- High Dose Setrusumab -> OL Setrusumab Selected Dose (Experimental): Single-blind setrusumab high dose during Phase 2 followed by open-label setrusumab
  During treatment and treatment extension periods, participants may receive supplementation with calcium and vitamin D to maintain normal values as directed by the treating physician
  Interventions: Biological: Setrusumab
- Setrusumab Selected Dose -> OL Setrusumab Selected Dose (Experimental): Double-blind setrusumab selected dose during Phase 3 followed by open-label setrusumab
  During treatment and treatment extension periods, participants may receive supplementation with calcium and vitamin D to maintain normal values as directed by the treating physician
  Interventions: Biological: Setrusumab
- Placebo -> OL Setrusumab Selected Dose (Placebo Comparator): Double-blind placebo during Phase 3 followed by open-label setrusumab
  During treatment and treatment extension periods, participants may receive supplementation with calcium and vitamin D to maintain normal values as directed by the treating physician
  Interventions: Biological: Setrusumab; Other: Placebo

INTERVENTIONS:
Biological: Setrusumab — A fully human sclerostin neutralizing monoclonal antibody (mAb) administered once a month (QM) via intravenous (IV) infusion
  Other Names: BPS804; UX143
Other: Placebo — A 5% dextrose/glucose solution administered QM via IV infusion
  Arms: Placebo -> OL Setrusumab Selected Dose

SUMMARY:
The primary objectives of the study are to identify a setrusumab dosing strategy in participants with OI and to evaluate the effect of setrusumab vs placebo on reduction in fracture rate.

DETAILED DESCRIPTION:
Participants in Phase 2 will be randomized 1:1 to receive low dose or high dose setrusumab. Phase 2 participants will continue receiving their assigned dose of setrusumab until all Phase 2 participants have completed the Month 6 study visit. After this point, Phase 2 participants will begin receiving the selected dosing strategy in the Phase 2 open-label Treatment Extension Period. Phase 3 participants will be randomized 2:1 to receive setrusumab or placebo during the double-blind treatment period. Phase 3 participants will transition to the open-label Treatment Extension Period after the end of the double-blind period. Participants in the Phase 2 and Phase 3 treatment extension periods will receive open-label setrusumab treatment for at least 12 months, and have the option to remain in the open-label treatment period until setrusumab is commercially available in their region. An optional substudy will be conducted in approximately 10 participants (≥ 8 years) consisting of a bone biopsy to investigate the impact of setrusumab on bone histomorphology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OI Type I, III, or IV as confirmed by identification of pathogenic or likely pathogenic genetic variants in COL1A1 or COL1A2. If a variant of uncertain significance is identified, then clinical presence of the expected phenotype can be used to confirm the diagnosis
* ≥ 1 fracture in the past 12 months, ≥ 2 fractures in the past 24 months or ≥ 1 tibia, femur or humerus fracture in the past 24 months
* Serum 25-hydroxyvitamin D ≥ 20 ng/mL at the Screening Visit. If 25-hydroxyvitamin D levels are below 20 ng/mL, 25-hydroxyvitamin D testing can repeated after a minimum of 14 days of vitamin D supplementation as directed by the treating physician
* Willing to not receive bisphosphonate therapy during the study
* From the period following informed consent to 60 days after the last dose of the study drug, females of childbearing potential and fertile males must consent to use highly effective contraception. If female, agree not to become pregnant. If male, agree not to father a child or donate sperm
* Willing and able to provide informed consent for subjects greater than or equal to 18 years of age, or provide assent (if possible) and have a legally authorized representative provide informed consent, after the nature of the study has been explained and prior to any research-related procedures
* Willing to provide access to medical records for the collection of radiographic data, fracture data, growth data, and disease history
* Must, in the opinion of the Investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule, and comply with the assessments

Exclusion Criteria:

* History of skeletal malignancies or bone metastases at any time
* History of neural foraminal stenosis (except if due to scoliosis)
* Clinical manifestations of Chiari malformation or basilar invagination. Presence of any other neurologic disease that has been unstable within past 2 years requires review by the Medical Monitor
* History of or uncontrolled concomitant diseases such as hypo/hyperparathyroidism, Paget's disease, abnormal thyroid function, thyroid disease or other endocrine disorders or conditions that could affect bone metabolism such as Stage IV/V renal disease
* Rickets or any skeletal condition (other than OI) leading to long-bone deformities and/or increased risk of fractures
* History of stroke, myocardial infarction, transient ischemic attack or angina.
* Hypocalcemia, defined as serum calcium levels below the age-adjusted normal limits after a ≥ 4 hour fast
* Estimated glomerular filtration rate ≤ 29 mL/min/1.73 m2
* Prior treatment with the following:

  1. Teriparatide, growth hormone, bone anabolic, or anti-resorptive medications (other than bisphosphonates) within 6 months of the first dose with study drug (Month 0)
  2. Denosumab within 24 months of Screening
  3. Romosozumab at any time
* Documented alcohol and/or drug abuse within 12 months prior to dosing or evidence of such abuse as indicated by the laboratory results during the Screening assessments
* Presence or history of any condition that, in the view of the Investigator, would interfere with participation, pose undue risk, or would confound interpretation of results
* Known hypersensitivity to setrusumab or excipients that, in the judgment of the Investigator, places the subject at increased risk for adverse effects
* History of external radiation therapy
* Pregnant or breastfeeding or planning to become pregnant (self or partner) at any time during the study
* Use of any investigational product or investigational medical device within 4 weeks or 5 half-lives of investigational drug (whichever is longer) prior to Screening, or during the study (per discretion of the Investigator in consultation with the Medical Monitor)
* Concurrent participation in another clinical study without prior approval from the Investigator in consultation with the Medical Monitor
* For Phase 2 Only: A history of bone surgery within the previous 6 months prior to Screening or planned bone surgery for the first 3 months of the study

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 183 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Percent Change in Serum Amino-terminal Propeptide of Type 1 Procollagen (P1NP) from Baseline at Month 1 | Baseline, Month 1
Phase 3: Annualized Rate of All Radiographically-Confirmed Fractures, Excluding Morphometric Vertebral Fractures and Fractures of the Fingers, Toes, Face, and Skull at the Primary Analysis | Up to Month 24

SECONDARY OUTCOMES:
Phase 2: Serum Setrusumab Concentration | From Predose up to Month 24
Phase 2: Baseline-Corrected Area Under the Effect Curve (AUEC) for Serum P1NP Over a 1 and 2-Month Period | Baseline, Up to Month 2
Phase 2: Percent Change from Baseline Over Time in Bone Turnover Marker: P1NP | Baseline, Up to Month 24
Phase 2: Percent Change from Baseline Over Time in Bone Turnover Marker: Osteocalcin (OCN) | Baseline, Up to Month 24
Phase 2: Change from Baseline in Dual Energy X-ray (DXA) Lumbar Spine Bone Mineral Density (BMD) Z-score Over Time | Baseline, Up to Month 24
Phase 2: Percent Change from Baseline in DXA Lumbar Spine BMD Over Time | Baseline, Up to Month 24
Phase 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Up to Month 24
Phase 2: Number of Participants With Anti-Setrusumab Binding and Neutralizing Antibodies | Up to Month 24
Phase 3: Annualized Rate of All Radiographically-Confirmed Fractures, Excluding Morphometric Vertebral Fractures, but Including Fractures of the Fingers, Toes, Face and Skull at the Primary Analysis | Up to Month 24
Phase 3: Annualized Rate of All Radiographically-Confirmed Fractures at the Primary Analysis | Up to Month 24
Phase 3: Change from Baseline in DXA Lumbar Spine BMD Z-score at the Primary Analysis | Baseline, up to Month 24
Phase 3: Change from Baseline in Pediatric Orthopedic Society of North America Pediatric Outcomes Data Collection Instrument (POSNA-PODCI) Sports/Physical Functioning Subscale Score for Pediatric Participants at the Primary Analysis | Baseline, up to Month 24
Phase 3: Proportion of Participants Experiencing New Radiographically Confirmed Fractures, Excluding Morphometric Vertebral Fractures and Fractures of the Fingers, Toes, Face, and Skull at the Primary Analysis | Up to Month 24
Phase 3: Change from Baseline in POSNA-PODCI Pain/Comfort Subscale Score for Pediatric Participants at the Primary Analysis | Baseline, Up to Month 24
Phase 3: Change from Baseline in 36-item Short Form Health Survey (SF-36) Physical Functioning Domain Scale for Adult Participants at the Primary Analysis | Baseline, Up to Month 24
Phase 3: Change from Baseline in SF-36 Bodily Pain (BP) Domain Scale for Adult Participants at the Primary Analysis | Baseline, Up to Month 24
Phase 3: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Up to Month 24
Phase 3: Number of Participants With Anti-Setrusumab Binding and Neutralizing Antibodies | Up to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Ultragenyx Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (44):
- United States (23):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Shriners Hospital for Children - Northern California, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Nemours/ Alfred i. duPoint Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Shriners Hospitals for Children - Chicago, Chicago, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center, Omaha, Nebraska
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Atrium Health Levine Children's Hospital, Charlotte, North Carolina
  - Nationwide Children's Hospital- Ohio State University College of Medicine, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - UW Health University Hospital, Madison, Wisconsin
- Australia (2):
  - Queensland Paediatric Endocrinology, South Brisbane, Queensland
  - Royal Children's Hospital, Melbourne
- Canada (4):
  - London Health Sciences Center, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - McGill University Health Centre, Montreal
  - University of Toronto- The Hospital for Sick Children (SickKids), Toronto
- Institut Imagine, Paris, France
- Germany (3):
  - University of Cologne, Cologne
  - Otto von Guericke University Magdeburg, Magdeburg
  - Musculoskeletal Center Würzburg, Würzburg
- Italy (3):
  - Istituto Ortopedico Rizzoli, Bologna
  - Azienda Ospedaliera Universitaria Policlinico Umberto I, Rome
  - Universita Degli Studi Di Verona, Verona
- Wilhelmina Children's Hospital, Utrecht, Netherlands
- Uniwersytet Medyczny w Lodzi - Klinika Endokrynologii i Chorob Metabolicznych, Lodz, Poland
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto, Porto
- Turkey (Türkiye) (2):
  - Gazi University, Ankara
  - Marmara University, Istanbul
- United Kingdom (2):
  - Royal Manchester Childrens Hospital, Manchester
  - Sheffield Children's NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Osteogenesis Imperfecta (OI) Research Study — https://www.ultraclinicaltrials.com/OI
- See also: Ultragenyx Transparency Commitment — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/